CLINICAL TRIAL: NCT05881304
Title: Switching Individuals in Treatment for Opioid Use Disorder Who Smoke Cigarettes to the SREC
Acronym: SWITCHED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joanna M. Streck, Ph.D., Assistant Professor in Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023p001364; K23DA056583 (NIH)
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Electronic Cigarette Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate SREC provision (iSREC) (Experimental): Those randomized to the iSREC group will be provided a free 8-week supply of standardized research e-cigarettes (SRECs) and asked to try to switch completely to the SREC.
  Interventions: Device: Standardized research e-cigarette (SREC)
- Delayed SREC provision waitlist control (WLC) (Active Comparator): Those in the WLC condition will receive SREC provision after an 8-week delay.
  Interventions: Device: Standardized research e-cigarette (SREC)

INTERVENTIONS:
Device: Standardized research e-cigarette (SREC) — Patients will be provided with NIDA's standardized research electronic cigarette (SREC) for 8-weeks and asked to attempt to substitute the SREC for combusted cigarettes during the 8 weeks. Participants will be randomized in a 1:1 ratio to 1 of 2 conditions for 8 weeks: 1) immediate standardized research e-cigarette provision (iSREC) or 2) delayed SREC provision waitlist control (WLC). Those randomized to the iSREC group will be provided a free 8-week supply of SRECs and asked to try to switch completely to the SREC. Those in the WLC condition will receive SREC provision after an 8-week delay.
  Other Names: SREC

SUMMARY:
The goal of this study is to conduct a pilot randomized waitlist-controlled trial to assess the feasibility, acceptability, and preliminary effects of substituting the NIDA standardized research e-cigarette (SREC) for combusted cigarettes in MOUD-TUD who are not ready to quit smoking. A waitlist controlled RCT using a mixed-methods sequential explanatory design will investigate the impact of SREC provision on: 1) tobacco use behavior (e.g., cigarettes per day [primary outcome], SREC use), 2) biomarkers (e.g., carbon monoxide, anabasine), 3) cigarette dependence and withdrawal, and 4) short-term health effects and tolerability (e.g., respiratory symptoms, substance use). In the proposed RCT, N=40 adults stable on MOUD with buprenorphine who report daily smoking recruited from MGH primary care practices will be randomly assigned to receive the SREC for 8 weeks, either immediately (iSREC), or after an 8-week delay (waitlist control [WLC]). They will be followed an additional 4 weeks after SREC provision ends (to 12 weeks in iSREC and 20 weeks in WLC).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age

  * Report daily cigarette smoking (>=10 cigarettes per day in the past week)
  * Not ready to quit smoking (not planning to quit in the next 30 days)
  * Willing to try e-cigarettes
  * In stable buprenorphine (BUP) treatment for opioid use disorder at an Massachusetts General Hospital-affiliated primary care clinic (in treatment for >=3 months without changes in BUP dose in the past 2 weeks and planning to remain on current BUP treatment for >=3 months).

Exclusion Criteria:

* Pregnant or breastfeeding
* Using non-cigarette nicotine or tobacco products (e.g., e-cigarettes, cigarillos) recently (>3 days in past 30 days)
* Report past 30-day use of behavioral or pharmacologic smoking cessation aids
* Deemed inappropriate for participation by their OUD provider
* Have an unstable psychiatric (e.g., past month suicidal ideation, active psychosis) or medical condition (e.g., life expectancy <1 year).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Cigarettes smoked per day | Baseline 2 to 8 weeks
  Change in cigarettes smoked per day (CPD) between randomized groups. Change in mean number of CPD in the past 7 days from Baseline 2 to Week 8 comparing between randomized groups (iSREC group vs. WLC).

SECONDARY OUTCOMES:
Study enrollment | Baseline
  Proportion of those screened identified as eligible. Proportion of those identified as eligible at screening who enroll in trial.
E-cigarette use during e-cigarette provision | During the 8 weeks of e-cigarette provision
  Mean days of e-cigarette use in past 7 days. 1) Number of days of e-cigarette use in past 7 days at Weeks 2, 4, 6, and 8 between randomized groups, and 2) number of days of e-cigarette use in the past 7 days in a pre-post analysis that combines randomized groups
Breath carbon monoxide | Baseline 1-Week 8
  Change in expired air carbon monoxide (CO)- during e-cigarette provision. Change in expired air CO (ppm) from Baseline to Week 8 between randomized groups.
Anabasine | Baseline 1-Week 8
  Change in anabasine - during e-cigarette provision. Change in urine anabasine level (ng/ml)from Baseline 1 to Week 8 between randomized groups.
Study completion | Baseline 2-12 weeks for iSREC (Baseline 2-20 weeks for WLC)
  Proportion of patients who complete the trial, defined as completing the final follow-up assessment (12 weeks for iSREC and 20 weeks for WLC) and >=50% of the study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna M Streck, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No